CLINICAL TRIAL: NCT07243392
Title: A Comparative Study on Effects of Steroid, Dextrose Prolotherapy, and Platelet-Rich Plasma Injections to Lessen Pain in Knee Osteoarthritis Patients
Brief Title: Effects of Steroid, Dextrose Prolotherapy, and Platelet-Rich Plasma Injections in Knee Joint OA Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lincoln University College (Other)
Responsible Party: Principal Investigator, Shahid sarwar, PhD Scholar, Lincoln University College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUC/CPGS/FOS/20250318/006
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthristis; Osteoarthritis, Knee; pain; steroids; Platelet-Rich Plasma; Injections, Intra-Articular; Regenerative Medicine.; Prolotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intra articular steroid injection (Experimental): Participants will receive intra-articular injections of corticosteroid such as methylprednisolone in order to reduce inflammation and manage pain.
  Interventions: Procedure: Intra articular steroid injection
- Intra articular PRP (Experimental): Participants will receive PRP, derived from the own blood of patient, which will be processed in laboratory to concentrate platelets containing growth factors to provide support in tissue repair.
  Interventions: Procedure: Intra articular PRP
- Intra articular dextrose prolotherapy (Experimental): Participants will receive dextrose prolotherapy injections, in which a hypertonic dextrose solution that is typically 25% will be injected into the knee joint in order to stimulate joint tissue regeneration.
  Interventions: Other: Intra articular dextrose prolotherapy

INTERVENTIONS:
Procedure: Intra articular steroid injection — Participants will receive intra-articular injections of corticosteroid such as methylprednisolone in order to reduce inflammation and manage pain.
  Arms: Intra articular steroid injection
Procedure: Intra articular PRP — Participants will receive PRP, derived from the own blood of patient, which will be processed in laboratory to concentrate platelets containing growth factors to provide support in tissue repair.
  Arms: Intra articular PRP
Other: Intra articular dextrose prolotherapy — Participants will receive dextrose prolotherapy injections, in which a hypertonic dextrose solution that is typically 25% will be injected into the knee joint in order to stimulate joint tissue regeneration.
  Arms: Intra articular dextrose prolotherapy

SUMMARY:
The novelty of thisstudy lies in its comparative assessment of three latest intra-articular injection therapies including steroid injections, dextrose prolotherapy, and PRP, for knee OA associated impairments, with a focus on long-term efficacy and safety profile. While prior studies may have assessed one or two of these treatments individually therefore this protocol is systematically designed.

DETAILED DESCRIPTION:
Osteo Arthritis (OA) is one of the chronic, Degenerative Joint Disease (DJD) categorized by the progressive loss of articular cartilage, leading to persistent joint pain, stiffness in the joints along with reduced mobility.

Knee OA has been documented as one of the principal causes of disability across the globe, with significantly higher incidence rate owing to physical trauma to joint, advancing age, obesity, and sedentary lifestyles etc. Management strategies for knee OA include following options, conservative management that include physiotherapy, adjunct therapies, pharmacological options and eventually surgical intervention such as knee replacements. Within the last few years, lots of focus has been placed on application of intra-articular injections for the knee joint which are reportedly found very effective in managing symptoms and altering the course of the disease without being too invasive. Among these, Corticosteroid Injections, Dextrose Prolotherapy and Platelet-Rich Plasma (PRP) injections stand out as the most common for the knee joint, each with its own unique mode of action and varying degree of effectiveness.

Corticosteroid intra-articular injections are known to be one of the most effective treatments. These injections provide relief in pain to joint inflammation targeting the synovial membrane through very potent anti-inflammatories injected directly into the joint.

Primary benefit of these injections is the speed of recovery with which pain is lessened and function of joint back to normal. A troublesome point of this approach is the pain relief time which is limited only a few weeks.

Literature has shown that excessive administration of corticosteroid intra-articular injections has resulted in the degradation of cartilage and narrowing of articular space, which could be antecedent to OA progression. As demonstrated in a randomized clinical trial, patients who were exposed to intra-articular triamcinolone at three-month intervals for a two-year period, experienced more cartilage volume loss over time, compared to placebo group participants highlighting the need for caution in regard to corticosteroids in the treatment of knee OA.

Dextrose prolotherapy is defined as a self augmenting injection therapy in w Dextrose prolotherapy is a unique approach with improvements in pain and function that persist over time, however, this approach likely takes a longer time for relief as compared to that of corticosteroids. Advantage of this therapeutic modality with PRP injections is that they are both anti inflammatory and regenerative in nature and thus, they provide both immediate and prolonged advantages excluding any significant risk to the patient.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria include patients aged 40-80 years, diagnosed with knee OA having Kellgren- Lawrence grades 2-4(Gelber, 2024) having history of persistent knee pain from at least last six months -

Patients Exclusion reporting with history of recent knee surgery, patients suffering from inflammatory joint diseases for example rheumatoid arthritis, having any active body infection, diabetic patients with de ranged HbA1c, pregnant and breast-feeding females will be excluded.:

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
NPRS | 9 months
  The Numeric Pain Rating Scale (NPRS) is a validated, self-reported measure used to assess pain intensity. Participants rate their current knee pain on a scale from 0 to 10, where 0 indicates "no pain" and 10 represents "worst imaginable pain." NPRS scores will be recorded at baseline and at designated follow-up intervals to evaluate the effectiveness of steroid, dextrose prolotherapy, and platelet-rich plasma injections in reducing pain among patients with knee osteoarthritis.
WOMAC | 9 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a validated, disease-specific, self-administered questionnaire used to assess pain, stiffness, and physical function in patients with knee and hip osteoarthritis. It consists of 24 items divided into three subscales:
  * Pain (5 items)
  * Stiffness (2 items)
  * Physical Function (17 items) Each item is rated on a Likert scale (0-4) or VAS (0-100 mm) depending on the version used. Higher scores indicate greater pain, stiffness, or functional limitation. WOMAC scores will be recorded at baseline and follow-up intervals to evaluate treatment efficacy across steroid, dextrose prolotherapy, and platelet-rich plasma injection groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Sarwar, Principal Investigator — Lincolin university college Malaysia
Locations (1):
- Health Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen KD, Thoma LM, Golightly YM. Epidemiology of osteoarthritis. Osteoarthritis Cartilage. 2022 Feb;30(2):184-195. doi: 10.1016/j.joca.2021.04.020. Epub 2021 Sep 14. PMID 34534661
- [Background] Arias-Vazquez PI, Tovilla-Zarate CA, Castillo-Avila RG, Legorreta-Ramirez BG, Lopez-Narvaez ML, Arcila-Novelo R, Gonzalez-Castro TB. Hypertonic Dextrose Prolotherapy, an Alternative to Intra-Articular Injections With Hyaluronic Acid in the Treatment of Knee Osteoarthritis: Systematic Review and Meta-analysis. Am J Phys Med Rehabil. 2022 Sep 1;101(9):816-825. doi: 10.1097/PHM.0000000000001918. Epub 2021 Nov 18. PMID 34740224
- [Background] Avdulaj, E. (2023). Comparative Analysis of Knee Replacement Surgery who follow up by Physical Therapy and Intra-articular Steroid Injections for Obese Patients. Albanian Journal of Trauma and Emergency Surgery, 7(2), 1300-1303.
- [Background] Berrigan WA, Bailowitz Z, Park A, Reddy A, Liu R, Lansdown D. A Greater Platelet Dose May Yield Better Clinical Outcomes for Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Systematic Review. Arthroscopy. 2025 Mar;41(3):809-817.e2. doi: 10.1016/j.arthro.2024.03.018. Epub 2024 Mar 19. PMID 38513880
- [Background] Cecerska-Heryc E, Goszka M, Serwin N, Roszak M, Grygorcewicz B, Heryc R, Dolegowska B. Applications of the regenerative capacity of platelets in modern medicine. Cytokine Growth Factor Rev. 2022 Apr;64:84-94. doi: 10.1016/j.cytogfr.2021.11.003. Epub 2021 Dec 2. PMID 34924312
- [Background] Gupta S, Paliczak A, Delgado D. Evidence-based indications of platelet-rich plasma therapy. Expert Rev Hematol. 2021 Jan;14(1):97-108. doi: 10.1080/17474086.2021.1860002. Epub 2020 Dec 17. PMID 33275468
- [Background] Ozturk MU, Baygutalp F. A comparative analysis of prolotherapy efficacy in patients with knee osteoarthritis across varied dextrose concentrations. Clin Rheumatol. 2023 Dec;42(12):3321-3331. doi: 10.1007/s10067-023-06723-4. Epub 2023 Aug 4. PMID 37540383